CLINICAL TRIAL: NCT00065312
Title: An Evaluation of an Oral Antidiabetic Agent for the Treatment of Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Purpose: Treatment
Other Study IDs: 5837; H7R-MC-GCBD
Record Dates: First submitted 2003-07-21; First posted 2003-07-22 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
Keywords: Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — naveglitazar

INTERVENTIONS:
Drug: naveglitazar

SUMMARY:
The purpose of this study is to determine if an investigational drug is safe and efficacious for poorly controlled type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 Diabetes for at least 3 months.
* Diabetes managed with diet and exercise alone or with either metformin or sulfonylurea alone as an adjunct to diet and exercise.
* Diabetes therapy must be unchanged for at least 3 months prior to screening.
* Females must be of non-childbearing potential (surgically sterilized or at least 1 year post-menopausal, as defined by cessation of menses). Female patients who are not surgically sterilized and who are less than or equal to 45 years should have their post-menopausal status confirmed by FSH greater that 30ng/mL at screening.

Exclusion Criteria:

* Current use of insulin or any antidiabetic agent other than a sulfonylurea agent or metformin.
* Current use of metformin or a sulfonylurea agent in combination.
* History of liver disease.
* History of unstable angina (as defined by the Braunwald system), myocardial infarction, or a coronary revascularization procedure within the past 6 months.
* Currently suspected carcinoma or history of carcinoma in the last 5 years, with the exception of excised superficial lesions such as basal cell carcinoma and squamous cell carcinoma of the skin.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (42):
- United States (42):
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Birmingham, Alabama
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Huntsville, Alabama
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Peoria, Arizona
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Tucson, Arizona
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Little Rock, Arkansas
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Bakersfield, California
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Pico Rivera, California
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), San Diego, California
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Santa Ana, California
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Denver, Colorado
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Waterbury, Connecticut
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), West Hartford, Connecticut
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Clearwater, Florida
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Kissimmee, Florida
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Ocala, Florida
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), St. Petersburg, Florida
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Decatur, Georgia
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Honolulu, Hawaii
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Orland Park, Illinois
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Peoria, Illinois
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Evansville, Indiana
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Wichita, Kansas
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Louisville, Kentucky
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Baltimore, Maryland
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Edina, Minnesota
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Minneapolis, Minnesota
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Endwell, New York
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Great Neck, New York
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Charlotte, North Carolina
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Fayetteville, North Carolina
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Oklahoma City, Oklahoma
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Eugene, Oregon
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Allentown, Pennsylvania
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Fleetwood, Pennsylvania
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Lansdale, Pennsylvania
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Philadelphia, Pennsylvania
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Mt. Pleasant, South Carolina
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), San Antonio, Texas
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Salt Lake City, Utah
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Lebanon, Virginia
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Renton, Washington
  - For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Spokane, Washington